CLINICAL TRIAL: NCT00955110
Title: An Exploratory, Single-Dose, Double-Blind, Randomized, Placebo-Controlled Crossover Study to Evaluate The Subjective and Objective Effects of Extended-Release Oxymorphone Compared to Controlled-Release Oxycodone in Healthy Non-Dependent Recreational Opioid Users
Brief Title: Study to Compare Oxymorphone Extended-Release (Opana ER) Versus Oxycodone Controlled-Release (Oxycontin)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: Kendle Early Stage - Toronto (Other)
Responsible Party: Sr. Director, Clinical R&D, Endo Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EN3202-402
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Opioid; Recreational; Oxymorphone; Oxycodone; Extended Release; Healthy NonDependent Recreational Opioid Users
MeSH Terms: interventions — Oxymorphone; Oxycodone; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Oxymorphone ER 15 mg (Experimental): 15mg
  Interventions: Drug: Oxymorphone ER; Drug: Hydromorphone
- Oxycodone CR 30 mg (Active Comparator): 30mg
  Interventions: Drug: Oxycodone CR; Drug: Hydromorphone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Hydromorphone
- Oxymorphone ER 30mg (Experimental): 30mg
  Interventions: Drug: Oxymorphone ER; Drug: Hydromorphone
- Oxycodone CR 60mg (Active Comparator): 60mg
  Interventions: Drug: Oxycodone CR; Drug: Hydromorphone

INTERVENTIONS:
Drug: Oxymorphone ER — 15mg or 30mg
  Other Names: Opana
  Arms: Oxymorphone ER 15 mg; Oxymorphone ER 30mg
Drug: Oxycodone CR — 30mg or 60mg
  Other Names: Oxycontin
  Arms: Oxycodone CR 30 mg; Oxycodone CR 60mg
Drug: Placebo — The placebo was a sugar pill.
  Arms: Placebo
Drug: Hydromorphone — 8 mg

SUMMARY:
The purpose of this study is to compare the subjective and objective effects of Oxymorphone ER (Opana ER) versus Oxycodone CR (Oxycontin).

ELIGIBILITY:
Inclusion Criteria:

* Recreational opioid use.
* At least 3 lifetime occasions of recreational use of an oral intact modified-release opioid product.
* BMI within range of 19.0 to 29.9 kg/m2, inclusive, minimum weight of 50.0 kg at screening and Day 0 of treatment period 1

Exclusion Criteria:

* Self-reported history of drug or alcohol dependence in the past 2 years or presence of drug or alcohol dependence in the past 12 months as defined by the DSM-IV, including subjects who have ever been in a drug rehabilitation program.
* Unwillingness or inability to abstain from recreational drug use as required for the study.
* History of acute asthma or other obstructive airway disease or any condition that may increase the risk for respiratory depression, judged as clinically significant by the investigator or designee.
* History of neurologic conditions such as convulsive disorders or severe head injury, judged as clinically significant by the investigator or qualified designee.
* History of Addison's disease, hypothyroidism, pancreatitis, prostatic hypertrophy, or urethral stricture.
* Use of non-prescription or prescription medications or natural health products within 7 days prior to first drug administration in the qualification phase and throughout the study, unless in the opinion of the investigator or designee, the product will not interfere with the study procedures or data integrity or compromise the safety of the subject.
* Uses of Monoamine oxidize inhibitors (MAOIs) within 14 days of first drug administration in the qualification phase and throughout the study.
* Current consumption of greater than 20 cigarettes (or 2 cigars) per day or inability to abstain from smoking (or use of any nicotine-containing sub stance) for at least 14 hours.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto, Ontario, Canada

REFERENCES:
- [Derived] Schoedel KA, McMorn S, Chakraborty B, Zerbe K, Sellers EM. Reduced cognitive and psychomotor impairment with extended-release oxymorphone versus controlled-release oxycodone. Pain Physician. 2010 Nov-Dec;13(6):561-73. PMID 21102969
- See also: Reduced Cognitive and Psychomotor Impairment with Extended-Release Oxymorphone Versus Controlled-Release Oxycodone — http://www.ncbi.nlm.nih.gov/pubmed/21102969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The period of recruitment was from 29 May 2009 (first subject enrolled) to 01 September 2009 (last subject completed).
Pre-assignment Details: A double-blind crossover qualification phase (hydromorphone 8 mg vs. placebo) was followed by a washout period and then randomization to a 5-period, 10-sequence crossover treatment phase. Approximately 40 qualified subjects were to be enrolled in the treatment phase in order to ensure that at least 30 subjects completed all 5 periods of the study.
Groups:
- All Subjects: Subjects enrolled were healthy non-dependent recreational opioid users. During the Treatment Phase, subjects were randomized to 1 of 10 treatment sequences, according to two 5 × 5 Williams squares. Subjects received single oral doses of each of the following 5 treatments, in a randomized, double-blind, crossover manner (1 capsule per treatment period): Placebo, Oxymorphone ER 15 mg, Oxymorphone ER 30 mg, Oxycodone CR 30 mg, and Oxycodone CR 60 mg.
  All participants did not necessarily receive the 5 drug interventions in the order reported as Milestones.
Period: Qualification Phase
Arm/Group | All Subjects
Started | 78
Completed | 54
Not Completed | 24
Not completed — Did not meet eligibility criteria | 24
Period: Treatment Phase
Arm/Group | All Subjects
Started | 41
Placebo | 38
Oxymorphone ER 15 mg | 37
Oxymorphone ER 30 mg | 38
Oxycodone CR 30 mg | 40
Oxycodone CR 60 mg | 40
Completed | 35
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Administrative reasons | 2
Not completed — Non-compliance with study restrictions | 1
Not completed — Withdrawn by physician pre-treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects Randomized to Treatment Phase: Forty one (41) qualified subjects were randomized into the treatment phase (Randomized population). Subjects were randomized to 1 of 10 treatment sequences, according to two 5 × 5 Williams squares. Subjects received single oral doses of each of the following 5 treatments, in a randomized, double-blind, crossover manner (1 capsule per treatment period): Placebo, Oxymorphone ER 15 mg, Oxymorphone ER 30 mg, Oxycodone CR 30 mg, and Oxycodone CR 60 mg.
Arm/Group | All Subjects Randomized to Treatment Phase
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 33
Region of Enrollment [Number; unit: participants]
  Canada | 41

OUTCOME MEASURES:

1. Primary Outcome: High VAS - Emax (mm)
Description: The High Visual Analog Scale (VAS) consisted of a horizontal line with a statement presented above the bar ("I am feeling high"). The ends of the line were marked with the descriptive anchors ("Definitely not" and "Definitely so"). Using a laptop computer, participants were instructed to click and drag the mouse to the appropriate position along the line, according to how they felt at that moment. Each scale was scored as an integer from 0 (Definitely not) to 100 (Definitely so), representing the position on the line.
Time Frame: High VAS was administered at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose.
Population: Per Protocol population: Subjects who received all 5 treatments and who had no major protocol deviations or other circumstances that would exclude them from the analysis. The pharmacokinetic and pharmacodynamic analyses were performed using the Per Protocol population. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Placebo: Subjects received a single oral dose (1 capsule) of placebo.
- Oxymorphone ER 15 mg: Subjects received a single oral dose (1 capsule) of Oxymorphone ER 15 mg.
- Oxymorphone ER 30 mg: Subjects received a single oral dose (1 capsule) of Oxymorphone ER 30 mg.
- Oxycodone CR 30 mg: Subjects received a single oral dose (1 capsule) of Oxycodone CR 30 mg.
- Oxycodone CR 60 mg: Subjects received a single oral dose (1 capsule) of Oxycodone CR 60 mg.
Arm/Group | Placebo | Oxymorphone ER 15 mg | Oxymorphone ER 30 mg | Oxycodone CR 30 mg | Oxycodone CR 60 mg
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35
mm | 23.1 (33.29) [33.29 to -16.0] | 30.6 (36.17) [-40.0 to -22.7] | 62.5 (33.22) [-19.0 to -10.6] | 81.4 (23.17) | 93.0 (12.94)
Statistical Analysis 1: Comparison: Oxymorphone ER 30 mg vs Oxycodone CR 60 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — A mixed-effect model for a crossover study was used, including treatment, period, treatment sequence and first-order carryover effect as fixed effects, pre-dose measurement as covariate, and subjects nested within treatment sequence as random effect; Least Square Means Difference = -28.8, 95% CI 2-sided [-41.6 to -16.0]
Statistical Analysis 2: Comparison: Oxymorphone ER 15 mg vs Oxycodone CR 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = -50.5, 95% CI 2-sided [-63.4 to -37.5]
Statistical Analysis 3: Comparison: Placebo vs Oxymorphone ER 15 mg; Test type: Superiority or Other; p = 0.395, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = 5.5, 95% CI 2-sided [-7.3 to 18.3]
Statistical Analysis 4: Comparison: Placebo vs Oxymorphone ER 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = 38.0, 95% CI 2-sided [25.2 to 50.8]
Statistical Analysis 5: Comparison: Placebo vs Oxycodone CR 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = 56.0, 95% CI 2-sided [43.1 to 68.9]
Statistical Analysis 6: Comparison: Placebo vs Oxycodone CR 60 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = 66.8, 95% CI 2-sided [53.9 to 79.7]

ADVERSE EVENTS:
Time Frame: AEs were documented in the eCRF and/or source documents, whether considered treatment-related or not related, throughout the study (ie, from first dose of study drug in the qualification phase to 30 days following the last dose of study drug).
Description: AEs were any new (or increased severity of) signs, symptoms, injury, or illness. Conditions existing prior to screening were recorded as the subject's medical history; events occurring from screening until first dose of study drug in the qualification phase were recorded as baseline signs and symptoms. AEs were reported for the safety population.
Groups:
- Treatment Phase Placebo: Identical placebo capsules using size AA Swedish orange capsules and microcrystalline cellulose.
- Treatment Phase Oxymorphone ER 15 mg: Single oral dose (1 capsule) of Oxymorphone HCl ER 15 mg (OPANA® ER), overencapsulated with size AA Swedish orange capsules with microcrystalline cellulose overfill.
- Treatment Phase Oxymorphone ER 30mg: Single oral dose (1 capsule) of Oxymorphone HCl ER 30 mg (OPANA® ER), overencapsulated with size AA Swedish orange capsules with microcrystalline cellulose overfill.
- Treatment Phase Oxycodone CR 30mg: Single oral dose (1 capsule) of Oxycodone HCl CR 30 mg (OxyContin®), overencapsulated with size AA Swedish orange capsules with microcrystalline cellulose overfill.
- Treatment Phase Oxycodone CR 60 mg: Single oral dose (1 capsule) of Oxycodone HCl CR 60 mg (OxyContin®), overencapsulated with size AA Swedish orange capsules with microcrystalline cellulose overfill.
Arm/Group | Treatment Phase Placebo | Treatment Phase Oxymorphone ER 15 mg | Treatment Phase Oxymorphone ER 30mg | Treatment Phase Oxycodone CR 30mg | Treatment Phase Oxycodone CR 60 mg
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37 | 0/38 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 13/38 | 22/37 | 28/38 | 35/40 | 39/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase Placebo (N=38) | Treatment Phase Oxymorphone ER 15 mg (N=37) | Treatment Phase Oxymorphone ER 30mg (N=38) | Treatment Phase Oxycodone CR 30mg (N=40) | Treatment Phase Oxycodone CR 60 mg (N=40)
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 6 | 18
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 9
Fatigue (General disorders) | 1 | 0 | 1 | 5 | 4
Feeling hot (General disorders) | 1 | 0 | 1 | 2 | 1
Feeling of relaxation (General disorders) | 3 | 2 | 3 | 3 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 4 | 2 | 7 | 8
Headache (Nervous system disorders) | 1 | 4 | 3 | 4 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
Sedation (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 7 | 8 | 10 | 12 | 13
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 2 | 1
Euphoric mood (Psychiatric disorders) | 2 | 9 | 20 | 27 | 37
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 7 | 8
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any analysis and/or publication of any data generated or arising from the study is not permitted without the prior written consent of Endo Pharmaceuticals Inc.